CLINICAL TRIAL: NCT02130778
Title: Natriuretic Effect of GLP-1 in Healthy Non Obese Subjects Followed by Oral Sodium Load: A Randomized, Placebo-controlled, Cross-over Study
Brief Title: Natriuretic Effect of GLP-1in Healthy Non Obese Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Maja Baretić, Maja Baretić, Clinical Hospital Centre Zagreb
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UHCZagreb
Record Dates: First submitted 2014-04-29; First posted 2014-05-05 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Sodium Excretion by Urination
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline infusion (Active Comparator): infusion of saline
  Interventions: Other: 500 ml 0.9% saline
- Saline infusion with GLP1 (Active Comparator): infusion of saline with GLP1
  Interventions: Drug: Synthetic GLP-1 (1.5 pmol/kg/min) dissolved in 500 ml 0.9% saline

INTERVENTIONS:
Drug: Synthetic GLP-1 (1.5 pmol/kg/min) dissolved in 500 ml 0.9% saline — infusion of synthetic GLP-1 (1.5 pmol/kg/min) saline
  Arms: Saline infusion with GLP1
Other: 500 ml 0.9% saline — infusion of saline
  Arms: Saline infusion

SUMMARY:
Adipose and diabetic patients have glomerular hyperfiltration and enhanced reabsorption of sodium in the kidney leading to fluid retention and hypertension. It is already known that obese mice (db/db) have salt retention and elevated intrarenal angiotensin II , and that the mechanism of the salt retention is similar to the one described in human beings. In experimental study from 2009 done by Hirata K and al., published in Biochemical and Biophysical Research Communications to both obese type 2 diabetic db/db mice and non-diabetic db/m mice hypertension was artificially induced (acute sodium-loading and angiotensin II-infusion). Two groups of mice were treated with exendin-4 or vehicle for 12 weeks. Obese type 2 diabetic db/db mice show high salt-sensitivity. Exendin-4 demonstrated anti-hypertensive effect in db/db mice and angiotensin II-infused mice, related to attenuation of high salt-sensitivity. That observation confirmed that exendin-4, a GLP-1 (Glucagon-like peptide-1) analogue, has extra-islet effect including the regulation of salt handling. More then ten years before mentioned observations the presence of GLP 1 receptors was confirmed all over the body, also in kidneys. In 2004 Gutzwiller published a study in Journal of Clinical Endocrinology and Metabolism that examined 15 healthy subjects and 16 obese men (mean body mass index, 36 kg/m2) in a double-blind, placebo-controlled, crossover study. After overnight fasting hypertonic saline was infuse followed by 3-h infusion of GLP-1. Intravenous infusions of GLP-1 enhanced sodium excretion, reduced H+ secretion, and reduced glomerular hyperfiltration in obese men. These findings suggest an action at the proximal renal tubule and a potential renoprotective effect. Two years later same author with colleagues published a new study in Digestion. In a part of new study he observed 8 volunteers. The protocol included intravenous salt load compared to the effect of an infusion of GLP-to isotonic saline (placebo). Extracellular volume expansion induced by an intravenous infusion of hypertonic saline was partially compensated by an increase in urinary sodium and water excretion with GLP-1. He explained that volume expansion was associated with increased renal perfusion, rise in glomerular filtration and the filtered sodium load. It was observed that GLP-1 is able to increase renal sodium excretion by 69% and urine volume by 86%. Considering all mentioned above it is obvious that GLP-1 have natriuretic effect, although its exact mechanism and clinical usefulness remain unclear. Both GLP1 analogues and inhibitors of DPP4 (dipeptidyl peptidase 4), elevate GLP1 level, and it would not be a surprise to observe similar natriuretic effects in the body. Since GLP 1 is a peptide given IV. or sc. there are on long-term studies that observe final possible effect no blood pressure, but GLP1 analogues and DPP4 inhibitors enhancing the incretin action demonstrate some antihypertensive properties. 2008 in a study done by Mistry GC and al., published in Journal of Clinical Pharmacology antihypertensive effect of sitagliptin was observed. In nineteen patients on stable treatment with antihypertensive agent(s) investigators found small but statistically significant reductions of 24-hour ambulatory blood pressure. There are no many definitive clues why the blood pressure should droop during any treatment that elevates serum GLP1. At the end of 2009 an analysis was published in American Journal of Hypertension, showing results from six trials including 2,171 subjects treated with exenatide for at least 6. Again, a significantly greater reduction in systolic blood pressure was confirmed, not giving an explanation why it happened so. Finally, Prof. Sjöholm from Karolinska institute Sweden published in Diabetes, obesity and metabolism a review concerning impact of GLP-1 on endothelial function. He mentioned again decreased blood pressure through improvements in diuresis and natriuresis, but he also added a new element, improved endothelial dysfunction through GLP-1 receptor-dependent pathway. Though there are many speculations, exact antihypertensive effects and water homeostasis of both GLP-1 itself, also of GLP1 analogues and DPP4 inhibitors is still unknown. Finally, recent review (Tanaka et all) from 2011 confirms mentioned speculations regarding natriuretic effect of GLP1, quote …" Incretin mimetics and DPP-IV inhibitors are a novel class of antihypertensive drugs with natriuretic properties. They can be used in the treatment of salt-sensitive hypertension, which is characterized by edema. The idea is to investigate the effect of GLP1 on diuresis/natriuresis compared with placebo in healthy non-obese people and to compare natriuresis with GLP-1, BNP (brain natriuretic peptide) and ADH (antidiuretic hormone) levels in serum.

DETAILED DESCRIPTION:
This is a cross-over study. Totally 15 participants will be randomized (or other number later determined by power test). The duration of the study is 9 days that will include 3 visits and screening visit before starting the study.

Screening (day -1) Inclusion criteria are fulfilled before approaching Visit 1 on screening. Participants are instructed do come next day fasting and to collect 24h of urine sample.

Visit 1 (day 1) Participant voluntarily agrees to participate by giving informed written consent. Baseline study assessment is going to be performed fasting: blood count and differential, blood chemistry (liver enzymes, sodium, potassium, calcium, phosphorus, magnesium, chloride, serum amorality, urea and creatinine, lipid panel including cholesterol, triglycerides, HDL and LDL cholesterol, coagulation, uric acid, glucose and insulin, renin activity, aldosterone, GLP1 level, T4 TSH-thyroid stimulating hormone, ADH, BNP) In the 24 h urine collection sodium, chloride and calcium excretion, osmolality, creatinine are going to be measured, glomerular filtration is going to be assessed by creatinine clearance, urin analysis with microscopy is going to be preformed, EKG, kidney ultrasound together with 24-h blood pressure monitor. HOMA2 (The Homeostasis Model Assessment ) index is calculated and a total body water percentage determinated via Bioelectrical Impedance Analysis. All samples of renin activity and aldosterone in a study are going to be taken while being in horizontal position at least for 3 hours. Participants are going to be randomized regarding the glucose tolerance test. First group it the one with fasting glucose 4,5 -5,7 mmol/L and at 2 hour OGTT (the amount of sodium in OGTT fluid used is 0,4 mg of sodium and 0,3 mg of chloride in 0,2 L of water) glucose level below 7.8 mmol/l. The other group is the one with fasting glucose from 5,7 to 7 mmol/l and/or at 2 hour OGTT glucose level form 7.8 mmol/l to 11,1 mmol/L (venous sample). Patients are instructed to come on the next day fasting again.

Visit 2 (day 2) is a next study assessment: 24-h blood pressure monitor is removed, after the overnight fast oral saline load is going to be given in a form of a standardized meal (soup) in a amount of 12 g of NaCl (average daily intake of salt in Croatia). The soup is going to be consumed in 30 minutes. Volunteers are going to be instructed to drink afterwards 1/2 L of water during next 1 h. Placebo in a form iv infusion of hypertonic saline is going to be given at a rate of 0.06 ml/kg/in and infused during 3 hours from beginning of oral sodium load. During 6 hours (from oral sodium load) urine is gong to be collected. Finally, blood samples are going to be drawn for glucose, insulin, sodium, potassium, serum osmolality, serum creatinine, renin activity, and aldosterone, BNP, ADH and GLP1 level after 3 and 6 hours. Sodium, chloride and calcium excretion, osmolality and creatinine are going to be measured in the urine after 3 hours. Patients are instructed to come again after 7 days fasting.

Visit 3 (day 9) after the overnight fast again oral sodium load is going to be given in a form of a standardized meal (soup) in a same amount as previous day and again consumed in 30 minutes, they are going to drink afterwards 1/2 L of water during next 1 h like pervious day. Synthetic GLP-1 (1.5 pmol/kg/min) dissolved in 500 ml 0.9% saline is going to be infused during 3 hours from beginning of oral sodium load. During 6 hours (from oral sodium load) urine is gong to be collected, blood samples are going to be drawn after 3 and 6 hours for the same analysis as in Visit 2, just like urine collection after 6 hours.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Participant is ≥18 and ≤70 years of age on day of signing informed consent
* Participant is a male, or a female who is unlikely to conceive, as indicated by at least one "yes" answer to the following questions:

  * Patient is a surgically sterilized female
  * Patient is a postmenopausal female ≥45 years of age with >2 years since last menses
  * Patient is a non-sterilized, premenopausal female and agrees to abstain from heterosexual activity or to use an adequate method of contraception ( Note: Acceptable methods of birth control are: hormonal contraceptive, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, or vasectomy)
* BMI ≥185 and ≤25
* Healthy as determined by:

  * Complete medical history, physical exam and
  * Standard 12-lead EKG
  * Complete blood count, blood chemistry , urinalysis with microscopy
  * Kidney USG
* Participant understands the study procedures, and risks involved with the study and voluntarily agree to participate by giving informed written consent.

Exclusion Criteria:• History of hypertension, diabetes (ADA guidelines), kidney disease

o Participant has impaired renal function defined as glomerular filtration lower than 90 calculated by Cockcroft-Gault formula and 24 creatinine, also by urinary protein excretion > 200 mg/day or continuing active urinary sediment

* History of myocardial infarction, cerebrovascular accident or transient ischemic attack
* History of malignancy within last 5 years
* Current febrile state
* Participant is pregnant or nursing woman
* Failure to give informed consent or comply with the protocol
* Participant has received treatment with an investigational drug within the prior 3 months or is otherwise participating in another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Evidence of the positive effect on natriuresis (level of sodium in urin sample) following the of GLP1 infusion | Within the 10 minutes after the infusion synthetic GLP-1 (1.5 pmol/kg/min) dissolved in 500 ml 0.9% saline

CONTACTS AND LOCATIONS:
Locations (2):
- Croatia (2):
  - University Hospital Centre, Zagreb
  - University hospital Centre Zagreb, Zagreb

REFERENCES:
- [Background] Gutzwiller JP, Tschopp S, Bock A, Zehnder CE, Huber AR, Kreyenbuehl M, Gutmann H, Drewe J, Henzen C, Goeke B, Beglinger C. Glucagon-like peptide 1 induces natriuresis in healthy subjects and in insulin-resistant obese men. J Clin Endocrinol Metab. 2004 Jun;89(6):3055-61. doi: 10.1210/jc.2003-031403. PMID 15181098
- [Derived] Baretic M, Kusec V, Pavlic-Renar I. Glucagon-Like Peptide-1 Infusion Suppresses Aldosterone Levels in Healthy Normal-Weight Individuals: Double-Blind, Placebo-Controlled Crossover Study. Diabetes Ther. 2018 Dec;9(6):2315-2324. doi: 10.1007/s13300-018-0517-y. Epub 2018 Oct 8. PMID 30298444